CLINICAL TRIAL: NCT06645613
Title: Precision TMS With Integrated Visualization and Analysis of Real-time E-field and EEG Source Imaging
Brief Title: TMS With Real-time E-field and EEG Source Imaging
Acronym: NetworkTMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lipeng Ning, PhD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024P001808
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers Only
Keywords: transcranial magnetic stimulation; magnetic resonance imaging; EEG

STUDY DESIGN:
Intervention Model Description: This is a sham-controlled cross-over study. The participants will take a random order of sham or real TMS stimulations.
Who Masked: Participant
Masking Description: A random order of sham and real stimulations will be applied to the participants. A sham TMS coil will be used in the sham stimulations to generate the same sound as the real TMS coil. Moreover, a pulsed electric current will be applied to the scalp of the participants, which generates a feeling similar to that of real stimulations. In this way, the participants will be blind to the stimulation status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham TMS coils will be applied to stimulate the brain targets. No magnetic field will be generated using the sham coil. It will play sounds similar to the true TMS stimulations with the pulsed weak electric current applied to the scalp to generate a similar feeling as in true stimulations.
  Interventions: Device: Transcranial Magnetic Stimulation Device
- Transcranial Magnetic Stimulation (Experimental): TMS with the intermittent theta burst stimulation protocol will be applied to the computed brain targets based on the MRI data of each participants.
  Interventions: Device: Transcranial Magnetic Stimulation Device

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation Device — Transcranial magnetic stimulation uses FDA-approved coils to generate varying magnetic fields in the brain of the participant and induce an electric field in the underlying brain tissue. The standard intermittent Theta Burst Stimulation (iTBS) TMS protocol will be applied in this study. The same coil can be applied to generate sham stimulations that only generate sound and stimulations to the scalp without stimulating the brain.

SUMMARY:
The goal of this study is to develop and validate an approach for accurate targeting and stimulation of brain networks using transcranial magnetic stimulation (TMS) using information from magnetic resonance imaging (MRI) data. This study requires two visits from each participant.

In the first visit, the participant will be scanned by MRI scanners to collect data from the brain.

Next, the data will be analyzed by the researcher to model the connections between different regions of the brain to determine the stimulation areas related to the so-called frontoparietal network.

In the second visit, the participants will take four TMS sessions with different types of stimulations applied to the computed targets and complete a computer-based task named multi-source interference task. Electroencephalogram (EEG) data will be collected during the TMS stimulations and tasks.

The main hypothesis is that applying TMS stimulations to the brain targets reduces the response time and response error in the tasks.

DETAILED DESCRIPTION:
The main goal of this study is to develop and validate an approach to target and stimulate brain networks using transcranial magnetic stimulation using information from magnetic resonance imaging (MRI).

Participants in this study will first be scanned using an MRI scanner to collect data from the brain. The MRI session will take about 40 minutes to acquire anatomical MRI, diffusion MRI, and resting-state functional MRI from the subjects.

Next, the researchers will analyze the MRI data to determine the stimulation areas of each participant. The method will provide two target areas in the brain, including an area in the left dorsolateral prefrontal cortex (DLPFC) and an area in the left inferior parietal lobule (IPL), which are involved in the frontoparietal network related to the executive control functions of the brain.

In the second visit, the participants will take TMS stimulations to the determined brain targets at DLPFC and IPL. The standard intermittent theta-burst (iTBS) protocol will be applied to the targets. To evaluate the effect of TMS stimulations, the participants will perform a computer-based task, named multi-source interference task (MSIT), before the TMS stimulation and another task after the TMS stimulations. The participants will click mouse buttons to respond to instructions in the tasks.

The response time and response error of the tasks will be the outcome measures of this study. The hypothesis is that applying TMS stimulations to the developed brain network targets reduces the response time and response error.

During the TMS stimulations and tasks, electroencephalogram (EEG) data will be collected from the participants. The EEG data, MRI data, and TMS-induced electric field maps will be analyzed and visualized using a software named SlicerTMS. However, the information shown in SlicerTMS will not be used to change the stimulation protocol in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 and less than 65 years.
2. Able to understand and give informed consent/assent.
3. No prior neuropsychiatric, neurological disorders, epilepsy, or seizures.
4. No metal implants.
5. Absent of lesions or tumors from MRI scans.

Exclusion Criteria:

1. The presence of a cardiac pacemaker or pacemaker wires.
2. Metallic particles in the eye.
3. Vascular clips in the head or previous neurosurgery.
4. Prosthetic heart valves.
5. Significant claustrophobia.
6. Non-fixed metallic particles (shrapnel).
7. Any magnetic metallic particles in the body.
8. Failure to assure non-pregnant status.
9. Failure to perform the task of lying still.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
choice reaction time (CRT) | 5 to 15 minutes right before and after each TMS session
  CRT is the time that the participant takes to click the mouse button in the computer-based Multi-Source Interference Task.

SECONDARY OUTCOMES:
response error | 5 to 15 minutes right before and after each TMS session
  The rate of incorrect response in the MSIT task.

CONTACTS AND LOCATIONS:
Locations (1):
- MGH at the Navy Yard, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No